CLINICAL TRIAL: NCT00135915
Title: Influence of Binge Drinking on Glucose Metabolism in Patients With Type 1 Diabetes - A Pilot Study
Status: Completed | Type: Observational
Sponsor: The Royal Bournemouth Hospital (Other)
Other Study IDs: BDEC ALC 1
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although there is no evidence that individuals with type 1 diabetes have a different approach to alcohol compared to the background population, nevertheless, its use does have implications for patients mainly because of the risk of hypoglycaemia unawareness. However, binge drinking has been implicated as a factor in the development of ketoacidosis and is probably under-recognised. The aim of this study is to examine the effect of binge drinking on glucose, insulin, counter-regulatory hormones and other metabolites in patients with type 1 diabetes. It is hoped that data from this project will be used to develop a larger study comparing different treatment regimens for patients using alcohol to reduce the risks of hyperglycaemia as well as hypoglycaemia.

DETAILED DESCRIPTION:
This is a randomised trial involving Type I diabetics who have had Type I diabetes >5 years. They will be using multiple daily injections of a basal insulin and a rapid acting component.Apart from insulin and oral contraceptive, none will be on regular medication. All will be regular consumers of modest amount of alcohol (Female - less than or equal to 14 units, males - less than or equal to 21 units). Each will participate in 2 studies. Subjects will be randomised either to white wine or an equivalent volume of alcohol-free wine.Outcome measures are the results of the effect of acute ingestion of alcohol on glucose levels and intermediate metabolites in subjects with Type I diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for > 5 years
* Use of multiple daily injections of a basal insulin and a rapid acting component
* Regular consumption of modest amounts of alcohol

Exclusion Criteria:

* Type 2 diabetes
* Type I diabetes < 5 years
* Excessive alcohol consumption
* Unstable diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females of at least 18 years of age who were diagnosed with Type 1 diabetes more than 5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-08; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, Doctor, Principal Investigator — The Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom